CLINICAL TRIAL: NCT07038109
Title: Effects of Progressive Muscle Relaxation on Depression, Anxiety, Stress, Future Attitudes, and Biopsychosocial Responses in Nursing Students: A Randomized Controlled Trial
Brief Title: Progressive Muscle Relaxation in Nursing Students: Effects on Psychological and Biopsychosocial Outcomes
Acronym: PRMNURSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ahsen Taştan Gürkan, Research Assistant, PhD in Nursing, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HEM-PGE-RCT-2024-TUBITAK2209-A; 1919B012327345 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey (TUBITAK))
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Depression; Anxiety; Stress, Psychological; Mental Health; Students, Nursing; Adaptation, Psychological; Psychophysiologic Disorders; Relaxation Therapy; Progressive Relaxation Exercise; Progressive Muscle Relaxation Exercise
Keywords: Progressive Muscle Relaxation; Psychological Intervention; Nursing Students; Mental Health Promotion; Stress Management; Depression; Anxiety; Psychological Stress; Biopsychosocial Response; Future Orientation; University Students; Randomized Controlled Trial; Relaxation Techniques; progressive relaxation exercise
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress, Psychological; Psychological Well-Being; Psychophysiologic Disorders | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: This study used a two-arm, parallel assignment design. Participants were randomly assigned to either the experimental group, which received progressive muscle relaxation exercises, or the control group, which received no intervention. A pretest-posttest design was used to assess outcomes.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded to their group allocation during the intervention process. The outcome assessor (statistician) was also blinded to group assignment during data analysis to reduce bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants in this group received progressive relaxation exercises (PRE) (Experimental): A structured progressive muscle relaxation program based on Jacobson's technique was implemented. The intervention lasted four weeks, with participants practicing three times per week in 45-minute sessions. The exercises were initially demonstrated in person by the researcher to ensure correct technique. Subsequently, participants followed pre-recorded audio instructions during each session to maintain consistency. The intervention aimed to reduce psychological symptoms and support biopsychosocial well-being in nursing students.
  Interventions: Other: Progressive relaxation exercise
- Control group (No Intervention): Participants in this group did not receive any behavioral or psychological intervention during the study period. They continued their normal academic activities without any additional support or guidance. No relaxation techniques or recordings were provided to this group. Data were collected at the same time points as the experimental group to ensure consistency in measurement.

INTERVENTIONS:
Other: Progressive relaxation exercise — The intervention was based on Jacobson's Progressive Muscle Relaxation (PMR) technique. Participants in the experimental group practiced PMR three times per week for four weeks. Each session lasted approximately 45 minutes and was conducted in a quiet environment. In the first session, the researcher provided face-to-face instruction. Subsequent sessions were guided by standardized audio recordings, and the participants were followed through scheduled online video calls. The intervention aimed to reduce depression, anxiety, and stress symptoms and to promote biopsychosocial well-being in nursing students.
  Other Names: progressive muscle relaxation; progressive muscle relaxation exercises; Progressive Relaxation Technique; Jacobson's Progressive Muscle Relaxation; Muscle Relaxation Exercise; Progressive Relaxation Training; Jacobson's progressive relaxation technique
  Arms: Participants in this group received progressive relaxation exercises (PRE)

SUMMARY:
This randomized controlled trial aims to investigate the effects of progressive muscle relaxation exercises (PMRE) on depression, anxiety, stress, future attitude, and biopsychosocial responses among nursing students. The study will be conducted between June 2024 and June 2025 at the Faculty of Health Sciences, Ondokuz Mayis University. Data collection will take place between January and March 2025. A total of 104 students will be randomly assigned to experimental and control groups. Data will be collected using the DASS-21, Future Orientation Scale, and the Biopsychosocial Response Scale for Nursing Students.

DETAILED DESCRIPTION:
Nursing students often face academic stress, emotional demands, and clinical responsibilities, which may lead to psychological difficulties such as depression, anxiety, stress, and concerns about their future. These problems can affect both their well-being and professional competence. Progressive muscle relaxation exercises (PMRE) are considered a beneficial method for reducing muscle tension, managing stress, and improving emotional regulation.

This randomized controlled trial is being conducted between June 2024 and June 2025 at the Faculty of Health Sciences, Ondokuz Mayis University. The data collection phase is scheduled from January to March 2025. A total of 104 nursing students will be randomly assigned to an experimental group (receiving PMRE) or a control group. A pretest-posttest design will be used. Measurement instruments include the Depression, Anxiety, and Stress Scale (DASS-21), the Future Orientation Scale, and the Biopsychosocial Response Scale for Nursing Students.

This study is supported by the Scientific and Technological Research Council of Turkey (TUBITAK), under the 2209-A University Students Research Projects Support Program.

ELIGIBILITY:
Inclusion Criteria:

* Being registered in the Department of Nursing
* Voluntary consent to participate in the study

Exclusion Criteria:

* Having joint or muscle pain, or any condition that may interfere with performing relaxation exercises
* Having a diagnosis of cancer or any chronic disease
* Having a psychiatric disorder that may interfere with obtaining valid results from the study (e.g., major depressive disorder, severe anxiety disorders, serious psychiatric conditions)
* Currently receiving antidepressant, anxiolytic, or similar psychiatric treatment
* Regular use of non-pharmacological methods such as yoga, psychotherapy, or similar practices

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Change in depression, anxiety, and stress levels measured by DASS-21 | Baseline and Week 4
  The Depression Anxiety Stress Scale - 21 (DASS-21) will be used to assess changes in psychological symptoms. It consists of three subscales measuring depression, anxiety, and stress. The scale will be administered at baseline (pre-test) and after the 4-week intervention (post-test).

SECONDARY OUTCOMES:
Change in future orientation levels measured by the Future Orientation Scale | Baseline and Week 4
  The Future Orientation Scale will be used to evaluate students' attitudes toward the future, including goal-setting, planning, and optimism. The scale will be administered before and after the intervention to detect changes.
Change in biopsychosocial response levels measured by the Biopsychosocial Response Scale for Nursing Students | Baseline and Week 4
  This scale measures students' emotional, physical, and social stress-related symptoms. It will be administered at baseline and after the intervention to assess changes in biopsychosocial well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to ethical restrictions and the scope of the study. The research was conducted as part of a TÜBİTAK 2209-A student project and approved only for academic use within the institution. No explicit consent or ethical approval was obtained for external data sharing.